CLINICAL TRIAL: NCT02507505
Title: A Randomized Controlled Trial of Regional Versus General Anesthesia for Promoting Independence After Hip Fracture
Brief Title: Regional Versus General Anesthesia for Promoting Independence After Hip Fracture
Acronym: REGAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 822632; PCORI-1406-18876 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, Conduction; Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regional Anesthesia (Active Comparator): Approximately half of the subjects will be randomized to the arm which receives Regional Anesthesia.
  Interventions: Procedure: Regional Anesthesia
- General Anesthesia (Active Comparator): Approximately half of the subjects will be randomized to the arm which receives General Anesthesia.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Regional Anesthesia — Regional anesthesia involves temporarily numbing parts of the body with nerve blocks. Spinal anesthesia is a type of regional anesthesia that uses medications injected into the fluid surrounding the spinal cord to temporarily numb the legs and lower abdomen. Spinal anesthesia is the most widely used type of regional anesthesia for hip fracture surgery. While intravenous sedation is typically used for comfort with spinal anesthesia, invasive airway interventions are not typically required.
  Other Names: Regional Block or Spinal Block
  Arms: Regional Anesthesia
Procedure: General Anesthesia — General anesthesia uses injected or inhaled medications to keep people unconscious during surgery. Since general anesthesia depresses breathing and impairs protective airway reflexes, invasive airway interventions such as breathing tube placement and mechanical ventilation are usually required.
  Other Names: General Endotracheal Anesthesia
  Arms: General Anesthesia

SUMMARY:
The purpose of this study is to find out if two types of standard care anesthesia are the same or if one is better for people who have hip fractures.

DETAILED DESCRIPTION:
Hip fracture is a clinical condition that involves a break in the femur (hip bone) near where it attaches to the pelvis. Hip fractures occur more than 300,000 times each year in the US and over 1.6 million times each year worldwide.

Over 90% of hip fractures occur in individuals aged 50 or older, most commonly resulting from low-energy traumatic injuries, such as falls from standing in the context of established osteoporosis, chronic illness, or disability. Surgical treatment, via fixation of the fractured bone or partial or total replacement of the hip joint, is indicated for all types of hip fractures and approximately 95% of hip fracture patients undergo surgery.

No evidence-based interventions now exist to improve functional outcomes after hip fracture surgery beyond the immediate postoperative period. Nearly all hip fracture patients require orthopedic surgery and anesthesia, making the anesthetic care episode a major opportunity to impact outcomes.

Spinal and general anesthesia represent the two standard care approaches to anesthesia for hip fracture surgery. Basic and clinical research has identified multiple plausible mechanisms by which spinal anesthesia may improve outcomes after hip fracture; nonetheless, major guidelines and systematic reviews have identified key evidence gaps and anesthesia care for hip fracture varies markedly in practice. While spinal and general anesthesia for hip fracture have been previously compared in retrospective studies and small randomized trials, much of the available prospective trial data is old and may not be reflective of current clinical practice.

REGAIN will be the first pragmatic multicenter prospective randomized trial of spinal versus general anesthesia for hip fracture surgery designed to evaluate the association of anesthesia technique with functional recovery after hip fracture. As such, it will fill critical evidence gaps to inform policy and practice.

Approximately 2,424 subjects will be enrolled (i.e. informed consent for participation will be obtained) in order to yield approximately 1,600 randomized patients. This estimate is based on an assumption that one in three patients (33%) who undergo consent prior to surgery will not be randomized on the day of surgery due to active clinical issues, timing of medication dosing, clinical assessments by treating physicians or the site Clinical Director or their designate, or patient withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or radiographically diagnosed intracapsular or extracapsular hip fracture
* Planned surgical treatment via hemiarthroplasty, total hip arthroplasty or appropriate fixation procedure
* Ability to walk 10 feet or across a room without human assistance before fracture

Exclusion Criteria:

* Planned concurrent surgery not amenable to spinal anesthesia
* Absolute contraindications to spinal anesthesia
* Periprosthetic fracture

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1848 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Neuman, MD, MSc, Principal Investigator — University of Pennsylvania
Locations (45):
- United States (38):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California Davis Medical Center, Sacramento, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - University of Florida Gainesville, Gainesville, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Florida Hospital, Winter Park, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospital & Clinics, Iowa City, Iowa
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Cooper University Hospital, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Rutgers-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - NYU-Winthrop Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Sacred Heart at RiverBend, Springfield, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Reading Hospital, Reading, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University Medical Center Brackenridge and Seton Medical Center Williamson, Austin, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Fairfax Medical Campus, Fairfax, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Simon Fraser Orthopaedic Fund - Royal Columbian Hospital, New Westminster, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Clapp JT, Dinh C, Hsu M, Neuman MD. Clinical reasoning in pragmatic trial randomization: a qualitative interview study. Trials. 2023 Jun 27;24(1):431. doi: 10.1186/s13063-023-07445-3. PMID 37365614
- [Derived] Neuman MD, Feng R, Ellenberg SS, Sieber F, Sessler DI, Magaziner J, Elkassabany N, Schwenk ES, Dillane D, Marcantonio ER, Menio D, Ayad S, Hassan M, Stone T, Papp S, Donegan D, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes R, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Tierney A, Gaskins LJ, Horan AD, Brown T, Dattilo J, Carson JL; REGAIN (Regional versus General Anesthesia for Promoting Independence after Hip Fracture) Investigators*; Looke T, Bent S, Franco-Mora A, Hedrick P, Newbern M, Tadros R, Pealer K, Vlassakov K, Buckley C, Gavin L, Gorbatov S, Gosnell J, Steen T, Vafai A, Zeballos J, Hruslinski J, Cardenas L, Berry A, Getchell J, Quercetti N, Bajracharya G, Billow D, Bloomfield M, Cuko E, Elyaderani MK, Hampton R, Honar H, Khoshknabi D, Kim D, Krahe D, Lew MM, Maheshwer CB, Niazi A, Saha P, Salih A, de Swart RJ, Volio A, Bolkus K, DeAngelis M, Dodson G, Gerritsen J, McEniry B, Mitrev L, Kwofie MK, Belliveau A, Bonazza F, Lloyd V, Panek I, Dabiri J, Chavez C, Craig J, Davidson T, Dietrichs C, Fleetwood C, Foley M, Getto C, Hailes S, Hermes S, Hooper A, Koener G, Kohls K, Law L, Lipp A, Losey A, Nelson W, Nieto M, Rogers P, Rutman S, Scales G, Sebastian B, Stanciu T, Lobel G, Giampiccolo M, Herman D, Kaufman M, Murphy B, Pau C, Puzio T, Veselsky M, Apostle K, Boyer D, Fan BC, Lee S, Lemke M, Merchant R, Moola F, Payne K, Perey B, Viskontas D, Poler M, D'Antonio P, O'Neill G, Abdullah A, Fish-Fuhrmann J, Giska M, Fidkowski C, Guthrie ST, Hakeos W, Hayes L, Hoegler J, Nowak K, Beck J, Cuff J, Gaski G, Haaser S, Holzman M, Malekzadeh AS, Ramsey L, Schulman J, Schwartzbach C, Azefor T, Davani A, Jaberi M, Masear C, Haider SB, Chungu C, Ebrahimi A, Fikry K, Marcantonio A, Shelvan A, Sanders D, Clarke C, Lawendy A, Schwartz G, Garg M, Kim J, Caruci J, Commeh E, Cuevas R, Cuff G, Franco L, Furgiuele D, Giuca M, Allman M, Barzideh O, Cossaro J, D'Arduini A, Farhi A, Gould J, Kafel J, Patel A, Peller A, Reshef H, Safur M, Toscano F, Tedore T, Akerman M, Brumberger E, Clark S, Friedlander R, Jegarl A, Lane J, Lyden JP, Mehta N, Murrell MT, Painter N, Ricci W, Sbrollini K, Sharma R, Steel PAD, Steinkamp M, Weinberg R, Wellman DS, Nader A, Fitzgerald P, Ritz M, Bryson G, Craig A, Farhat C, Gammon B, Gofton W, Harris N, Lalonde K, Liew A, Meulenkamp B, Sonnenburg K, Wai E, Wilkin G, Troxell K, Alderfer ME, Brannen J, Cupitt C, Gerhart S, McLin R, Sheidy J, Yurick K, Chen F, Dragert K, Kiss G, Malveaux H, McCloskey D, Mellender S, Mungekar SS, Noveck H, Sagebien C, Biby L, McKelvy G, Richards A, Abola R, Ayala B, Halper D, Mavarez A, Rizwan S, Choi S, Awad I, Flynn B, Henry P, Jenkinson R, Kaustov L, Lappin E, McHardy P, Singh A, Donnelly J, Gonzalez M, Haydel C, Livelsberger J, Pazionis T, Slattery B, Vazquez-Trejo M, Baratta J, Cirullo M, Deiling B, Deschamps L, Glick M, Katz D, Krieg J, Lessin J, Mojica J, Torjman M, Jin R, Salpeter MJ, Powell M, Simmons J, Lawson P, Kukreja P, Graves S, Sturdivant A, Bryant A, Crump SJ, Verrier M, Green J, Menon M, Applegate R, Arias A, Pineiro N, Uppington J, Wolinsky P, Gunnett A, Hagen J, Harris S, Hollen K, Holloway B, Horodyski MB, Pogue T, Ramani R, Smith C, Woods A, Warrick M, Flynn K, Mongan P, Ranganath Y, Fernholz S, Ingersoll-Weng E, Marian A, Seering M, Sibenaller Z, Stout L, Wagner A, Walter A, Wong C, Orwig D, Goud M, Helker C, Mezenghie L, Montgomery B, Preston P, Schwartz JS, Weber R, Fleisher LA, Mehta S, Stephens-Shields AJ, Dinh C, Chelly JE, Goel S, Goncz W, Kawabe T, Khetarpal S, Monroe A, Shick V, Breidenstein M, Dominick T, Friend A, Mathews D, Lennertz R, Sanders R, Akere H, Balweg T, Bo A, Doro C, Goodspeed D, Lang G, Parker M, Rettammel A, Roth M, White M, Whiting P, Allen BFS, Baker T, Craven D, McEvoy M, Turnbo T, Kates S, Morgan M, Willoughby T, Weigel W, Auyong D, Fox E, Welsh T, Cusson B, Dobson S, Edwards C, Harris L, Henshaw D, Johnson K, McKinney G, Miller S, Reynolds J, Segal BS, Turner J, VanEenenaam D, Weller R, Lei J, Treggiari M, Akhtar S, Blessing M, Johnson C, Kampp M, Kunze K, O'Connor M, Looke T, Tadros R, Vlassakov K, Cardenas L, Bolkus K, Mitrev L, Kwofie MK, Dabiri J, Lobel G, Poler M, Giska M, Sanders D, Schwartz G, Giuca M, Tedore T, Nader A, Bryson G, Troxell K, Kiss G, Choi S, Powell M, Applegate R, Warrick M, Ranganath Y, Chelly JE, Lennertz R, Sanders R, Allen BFS, Kates S, Weigel W, Li J, Wijeysundera DN, Kheterpal S, Moore RH, Smith AK, Tosi LL, Looke T, Mehta S, Fleisher L, Hruslinski J, Ramsey L, Langlois C, Mezenghie L, Montgomery B, Oduwole S, Rose T; REGAIN (Regional versus General Anesthesia for Promoting Independence after Hip Fracture) Investigators. Pain, Analgesic Use, and Patient Satisfaction With Spinal Versus General Anesthesia for Hip Fracture Surgery : A Randomized Clinical Trial. Ann Intern Med. 2022 Jul;175(7):952-960. doi: 10.7326/M22-0320. Epub 2022 Jun 14. PMID 35696684
- [Derived] Neuman MD, Feng R, Carson JL, Gaskins LJ, Dillane D, Sessler DI, Sieber F, Magaziner J, Marcantonio ER, Mehta S, Menio D, Ayad S, Stone T, Papp S, Schwenk ES, Elkassabany N, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes RA, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Giska M, Ranganath Y, Tedore T, Choi S, Li J, Kwofie MK, Nader A, Sanders RD, Allen BFS, Vlassakov K, Kates S, Fleisher LA, Dattilo J, Tierney A, Stephens-Shields AJ, Ellenberg SS; REGAIN Investigators. Spinal Anesthesia or General Anesthesia for Hip Surgery in Older Adults. N Engl J Med. 2021 Nov 25;385(22):2025-2035. doi: 10.1056/NEJMoa2113514. Epub 2021 Oct 9. PMID 34623788
- [Derived] Neuman MD, Gaskins LJ, Ziolek T; REGAIN Investigators. Time to institutional review board approval with local versus central review in a multicenter pragmatic trial. Clin Trials. 2018 Feb;15(1):107-111. doi: 10.1177/1740774517735536. Epub 2017 Oct 6. PMID 28982261
- [Derived] Neuman MD, Ellenberg SS, Sieber FE, Magaziner JS, Feng R, Carson JL; REGAIN Investigators. Regional versus General Anesthesia for Promoting Independence after Hip Fracture (REGAIN): protocol for a pragmatic, international multicentre trial. BMJ Open. 2016 Nov 15;6(11):e013473. doi: 10.1136/bmjopen-2016-013473. PMID 27852723

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1848 participants who provided informed consent, 248 withdrew consent prior to randomization; 1600 participants were randomly assigned to a treatment group and continued in the study.
Period: Overall Study
Arm/Group | Regional Anesthesia | General Anesthesia
Started | 795 | 805
Completed | 712 | 733
Not Completed | 83 | 72
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Participant unable to be contacted within 60-day interview window | 56 | 44
Not completed — Participant contacted but walking status was unknown | 14 | 16
Not completed — Death before receipt of anesthesia | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regional Anesthesia | General Anesthesia | Total
Number analyzed (Participants) | 795 | 805 | 1600
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (10.7) | 78.4 (10.6) | 78.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 537 | 535 | 1072
  Male | 258 | 270 | 528
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race was reported by patients or their proxies; number analyzed is the number of participants who provided data for this Baseline Measure.
  Participants
    White: number analyzed (Participants) | 762 | 774 | 1536
    White | 683 | 691 | 1374
    Black: number analyzed (Participants) | 762 | 774 | 1536
    Black | 55 | 67 | 122
    Other or more than one race: number analyzed (Participants) | 762 | 774 | 1536
    Other or more than one race | 24 | 16 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Ethnicity was reported by patients or their proxies. Data missing for some participants.
  Participants
    Hispanic ethnic group: number analyzed (Participants) | 750 | 763 | 1513
    Hispanic ethnic group | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  Canada | 210 | 212 | 422
  United States | 585 | 593 | 1178
3D-CAM Assessment for Delirium [Count of Participants; unit: Participants] — 3D-CAM Assessment positive for delirium prior to randomization Population: Only participants with completed baseline 3D-CAM assessments are included.
  Participants
    number analyzed (Participants) | 746 | 753 | 1499
    (all) | 96 | 104 | 200

OUTCOME MEASURES:

1. Primary Outcome: Death or Inability to Walk 10 Feet or Across a Room Without Human Assistance
Description: Will be assessed via telephone interview
Time Frame: Approximately 60 days after Randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 712 | 733
Participants | 132 | 132

2. Secondary Outcome: Overall Health and Disability
Description: Will be assessed via the 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0). The 12-item WHODAS 2.0 scale measures disability in six functional domains (cognition, mobility, self-care, social interaction, life activities, and community participation). Scores range from 0 to 100, with lower scores indicating lower degrees of disability.
Time Frame: Approximately 60, 180, and 365 days after randomization
Population: Patients providing data at each time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 280 | 276
score on a scale
  60-day outcome: number analyzed (Participants) | 225 | 241
  60-day outcome | 22.7 [8.3 to 43.2] | 18.2 [6.3 to 31.8]
  180-day outcome: number analyzed (Participants) | 249 | 274
  180-day outcome | 10.4 [2.3 to 27.1] | 10.4 [2.1 to 27.3]
  365-day outcome | 10.4 [2.1 to 29.2] | 8.3 [0 to 22.9]

3. Secondary Outcome: Ability to Return to Home
Description: Will be assessed via telephone interview. Measure assessed as death or new transition to nursing home residence at each time point.
Time Frame: Approximately 60, 180, and 365 days after randomization
Population: This outcome was assessed among patients who were not admitted from a nursing home, rehabilitation facility, or acute care hospital. Denominator includes all known decedents at each time point, plus survivors providing information on location of residence at the time of study interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 613 | 625
Participants
  60-day outcomes | 108 | 114
  180-day outcomes: number analyzed (Participants) | 594 | 597
  180-day outcomes | 103 | 90
  365-day outcomes: number analyzed (Participants) | 584 | 572
  365-day outcomes | 119 | 116

4. Secondary Outcome: Chronic Pain
Description: Will be assessed via the Numeric Rating Scale (NRS) and the need for prescription medications as evaluated during telephone interview. NRS values range from 0 to 10, with higher values indicating greater pain.
Time Frame: Approximately 60, 180, and 365 days after randomization
Population: Numbers differ across rows due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 315 | 320
units on a scale
  60-day measure | 4.5 (3.2) | 4.2 (3.2)
  180-day measure: number analyzed (Participants) | 284 | 302
  180-day measure | 3.5 (3.3) | 3.4 (3.3)
  365-day measure: number analyzed (Participants) | 266 | 275
  365-day measure | 3.1 (3.2) | 3.2 (3.3)

5. Secondary Outcome: Cognitive Function
Description: Will be assessed via Short Blessed Test (SBT); SBT values range from 0 to 28, with higher scores indicating greater degrees of cognitive impairment.
Time Frame: Baseline and approximately 60, 180, and 365 days after randomization
Population: Numbers differ across rows due to missing data
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 246 | 243
units on a scale
  60 day measure | 2 [0 to 5] | 2 [0 to 6]
  180 day measure: number analyzed (Participants) | 219 | 242
  180 day measure | 2 [0 to 6] | 2 [0 to 6]
  365 day measure: number analyzed (Participants) | 207 | 218
  365 day measure | 2 [0 to 4] | 2 [0 to 4]

6. Secondary Outcome: All-cause Mortality
Description: Will be assessed via telephone interview and National Death Index (NDI) search
Time Frame: Approximately 60, 180, and 365 days after randomization
Population: All enrolled patients who had not withdrawn or been lost to follow up a given study time point
Measure: Number; unit: participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 768 | 784
participants
  60-day outcomes | 30 | 32
  180-day outcomes: number analyzed (Participants) | 738 | 751
  180-day outcomes | 69 | 63
  365-day outcomes: number analyzed (Participants) | 714 | 712
  365-day outcomes | 98 | 92

7. Secondary Outcome: Need for Assistive Devices for Walking
Description: Will be assessed via telephone interview
Time Frame: Approximately 60, 180, and 365 days after randomization
Population: 60-day outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 672 | 694
Participants
  60 day outcomes: number analyzed (Participants) | 672 | 693
  60 day outcomes | 403 | 397
  180 day outcomes: number analyzed (Participants) | 614 | 638
  180 day outcomes | 231 | 231
  365 day outcomes: number analyzed (Participants) | 573 | 578
  365 day outcomes | 196 | 193

8. Secondary Outcome: Acute Postoperative Pain
Description: Will be assessed via in-person interview using numeric rating scale (NRS). NRS values range from 0 to 10, with greater values indicating worse pain.
Time Frame: Before surgery and daily through postoperative day 3 or day of discharge, whichever occurs first
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 706 | 722
units on a scale
  Postoperative day 1 | 7.9 (2.6) | 7.6 (2.8)
  Postoperative day 2 | 7.1 (2.7) | 7.1 (2.8)
  Postoperative day 3 | 6.8 (2.9) | 6.6 (3.0)

9. Secondary Outcome: Satisfaction With Care
Description: Will be assessed via Bauer Patient Satisfaction Questionnaire. Data reported here corresponds to a response of "dissatisfied" or "very dissatisfied" to one or more of 5 Bauer questionnaire items assessing the following domains: information given by anesthesiologist before surgery; waking up from anesthesia; pain therapy after surgery; treatment of nausea and vomiting after surgery; care provided by department of anesthesia in general.
Time Frame: Postoperative day 3 or day of discharge, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 647 | 661
Participants | 85 | 97

10. Secondary Outcome: Postoperative Delirium
Description: Will be assessed via 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) assessment tool. Any positive 3D-CAM screen over the first 3 postoperative days in a patient with a negative pre-randomization screen was counted as a case of incident delirium.
Time Frame: Baseline and daily through postoperative day 3 or day of discharge, whichever occurs first
Population: This outcome was assessed only among patients who had a negative 3D-CAM assessment for delirium before randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 633 | 629
Participants | 130 | 124

11. Secondary Outcome: Inpatient Mortality
Description: Will be assessed via medical chart review. Data reported here on inpatient mortality.
Time Frame: During initial hospitalization until day of discharge or 30 days after randomization, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 782 | 790
Participants | 5 | 13

12. Secondary Outcome: Major Inpatient Morbidity
Description: Indicates occurrence of any of 12 complications based on medical record review: Myocardial infarction; Nonfatal cardiac arrest; Stroke; Pneumonia; Pulmonary edema; Pulmonary embolism; Unplanned postoperative intubation; Surgical-site infection; Urinary tract infection; Any return to the operating room; Critical care admission; Acute kidney injury.
Time Frame: During initial hospitalization until day of discharge or 30 days after randomization, whichever occurs first
Measure: Count of Participants; unit: Participants
Arm/Group | Regional Anesthesia | General Anesthesia
Number analyzed (Participants) | 795 | 805
Participants | 98 | 120

ADVERSE EVENTS:
Time Frame: Adverse data were collected for up to one year post-randomization.
Arm/Group | Regional Anesthesia | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 98/795 | 92/805
Serious Adverse Events (participants affected / at risk) | 255/795 | 242/805
Other Adverse Events (participants affected / at risk) | 278/795 | 286/805
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regional Anesthesia (N=795) | General Anesthesia (N=805)
Anemia (Blood and lymphatic system disorders) | 52 | 48
Anemia associated with other specified nutritional deficiency (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3
Leukopenia NOS (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 4
Atrial flutter (Cardiac disorders) | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 4 | 5
Cardiogenic shock (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 6 | 1
Heart failure (Cardiac disorders) | 6 | 7
Myocardial infarction (Cardiac disorders) | 10 | 9
Sinus tachycardia (Cardiac disorders) | 3 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Femoral anteversion (Congenital, familial and genetic disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 5
Epigastric pain (Gastrointestinal disorders) | 1 | 0
Esophageal obstruction (Gastrointestinal disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 2 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
GI bleed (Gastrointestinal disorders) | 1 | 1
GI hemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatal hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Death (General disorders) | 0 | 1
Death NOS (General disorders) | 62 | 67
Edema limbs (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 4 | 3
Flu like symptoms (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 2
Multi-organ failure (General disorders) | 0 | 1
Pain (General disorders) | 4 | 4
Weakness (General disorders) | 1 | 0
Weakness generalized (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Ischemic hepatitis (Hepatobiliary disorders) | 0 | 1
Obstructive jaundice (Hepatobiliary disorders) | 1 | 0
Acute diverticulitis (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Bone infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Cystitis bacterial (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 1 | 0
Infection NOS (Infections and infestations) | 1 | 0
Joint infection (Infections and infestations) | 2 | 1
Kidney infection (Infections and infestations) | 1 | 0
Klebsiella pneumonia (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Post procedural pneumonia (Infections and infestations) | 9 | 9
Post procedural site wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 10 | 4
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 20 | 16
Wound infection (Infections and infestations) | 3 | 2
Acute kidney injury (Injury, poisoning and procedural complications) | 13 | 18
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 13 | 25
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 9 | 10
Fractured radial head (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 5 | 9
Laceration of head (Injury, poisoning and procedural complications) | 0 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 3
Post procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 | 2
Post procedural stroke (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Biopsy of lymph node (Investigations) | 1 | 0
Cardiac troponin I increased (Investigations) | 2 | 4
Cardiac troponin T increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Crossmatch incompatible (Investigations) | 1 | 0
Cystoscopy (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
INR increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Supratherapeutic INR (Investigations) | 1 | 0
Troponin increased (Investigations) | 4 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 4
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Other severe protein-calorie malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Nonunion of fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant liver tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urothelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 8 | 2
Intracranial hemorrhage (Nervous system disorders) | 3 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Stroke (Nervous system disorders) | 11 | 8
Syncope (Nervous system disorders) | 4 | 2
Syncope vasovagal (Nervous system disorders) | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 0 | 1
Trigeminal nerve disorder (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 5 | 3
Delirium (Psychiatric disorders) | 10 | 12
Delusions (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 2
Psychiatric disorder NOS (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 3
Acute renal failure (Renal and urinary disorders) | 5 | 8
Bladder perforation (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Kidney failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 4
Urinary tract obstruction (Renal and urinary disorders) | 3 | 1
Urine discoloration (Renal and urinary disorders) | 1 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hospital acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Lung cancer stage unspecified (excl metastatic tumours to lung) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4
SOB (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Arthroplasty of hip (Surgical and medical procedures) | 0 | 1
Bladder neoplasm surgery (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 | 1
Fracture repair (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Hospitalization (Surgical and medical procedures) | 0 | 1
Joint prosthesis replacement (Surgical and medical procedures) | 0 | 2
Lumbar laminectomy (Surgical and medical procedures) | 1 | 0
Revision of hip arthroplasty (Surgical and medical procedures) | 1 | 0
Total knee replacement (Surgical and medical procedures) | 1 | 0
Transfusion (Surgical and medical procedures) | 27 | 29
Wound debridement (Surgical and medical procedures) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Arterial thromboembolism (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 17 | 12
Hypovolemic shock (Vascular disorders) | 1 | 0
Peripheral ischemia (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 10 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regional Anesthesia (N=795) | General Anesthesia (N=805)
Anemia (Blood and lymphatic system disorders) | 73 | 75
Anemia iron deficiency (Blood and lymphatic system disorders) | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 | 1
Hypoplastic marrow (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 10 | 10
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Aortic valve disease (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 4
Chest pain - cardiac (Cardiac disorders) | 9 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 3 | 2
Heart failure, congestive (Cardiac disorders) | 0 | 1
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 13 | 7
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Urachal abnormality (Congenital, familial and genetic disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Euthyroid sick syndrome (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 3
Glaucoma (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 10 | 12
Diarrhea (Gastrointestinal disorders) | 3 | 6
Dry mouth (Gastrointestinal disorders) | 2 | 2
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 6
Emesis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 26 | 25
Pain anal (Gastrointestinal disorders) | 0 | 1
Regional ileitis aggravated (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 10
Chills (General disorders) | 7 | 3
Death from natural causes (General disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 4
Fatigue (General disorders) | 4 | 1
Fever (General disorders) | 20 | 17
Fever of unknown origin (General disorders) | 1 | 0
Foggy feeling in head (General disorders) | 1 | 0
Generalized edema (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 2
Pain (General disorders) | 20 | 14
Pyrexia (General disorders) | 1 | 0
Thirst (General disorders) | 13 | 12
Weakness (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Bacterial infection due to staphylococcus aureus (Infections and infestations) | 1 | 0
Bladder infection (Infections and infestations) | 2 | 0
Helicobacter pylori infection (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Post procedural pneumonia (Infections and infestations) | 1 | 4
Skin infection (Infections and infestations) | 1 | 0
Thrush (Infections and infestations) | 1 | 1
UTI (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 30 | 25
Vaginal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 2 | 0
Acute kidney injury (Injury, poisoning and procedural complications) | 7 | 10
Bruising (Injury, poisoning and procedural complications) | 1 | 1
Contusion of knee (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 7
Fracture (Injury, poisoning and procedural complications) | 5 | 3
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Lithium toxicity (Injury, poisoning and procedural complications) | 1 | 0
Meniscus tear (Injury, poisoning and procedural complications) | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1
Post procedural stroke (Injury, poisoning and procedural complications) | 1 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Tear of medial cartilage or meniscus of knee, current (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 1
Bilirubin increased (Investigations) | 1 | 0
BUN increased (Investigations) | 1 | 0
Cardiac troponin I increased (Investigations) | 1 | 1
Cardiac troponin T increased (Investigations) | 1 | 2
INR increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 3 | 3
Troponin increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyslipidemia (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3
Hypokalemic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 14 | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 4
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Other and unspecified protein-calorie malnutrition (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Baker's cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Limbs stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in heel (Musculoskeletal and connective tissue disorders) | 0 | 1
Ruptured intervertebral disc (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral hemorrhage (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 9 | 4
Dizziness exertional (Nervous system disorders) | 0 | 1
Drowsiness (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 6 | 4
Headache (Nervous system disorders) | 6 | 1
Lethargy (Nervous system disorders) | 1 | 2
Numbness of lower extremities (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 1
Seizure (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 10 | 10
Spasticity (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 4
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 2 | 2
Alcoholic withdrawal symptoms (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 3
Combative reaction (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 9 | 15
Delirium (Psychiatric disorders) | 15 | 22
Depression (Psychiatric disorders) | 2 | 0
Hallucinations (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Somatization disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2
Acute renal failure (Renal and urinary disorders) | 6 | 4
Chronic kidney disease (Renal and urinary disorders) | 1 | 2
Hematuria (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Retention urinary (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 16 | 22
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pressure ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 | 3
Blood transfusion (Surgical and medical procedures) | 2 | 0
Breast reconstruction (Surgical and medical procedures) | 0 | 1
Fracture treatment (Surgical and medical procedures) | 1 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Hip replacement (Surgical and medical procedures) | 0 | 1
Hip surgery (Surgical and medical procedures) | 0 | 1
Packed red blood cell transfusion (Surgical and medical procedures) | 2 | 2
Prostate transurethral resection (Surgical and medical procedures) | 0 | 1
Removal of other matter from skin or subcutaneous tissue (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Total knee replacement (Surgical and medical procedures) | 1 | 0
Transfusion (Surgical and medical procedures) | 44 | 59
DVT (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 8 | 6
Hypotension (Vascular disorders) | 22 | 17
Orthostatic hypotension (Vascular disorders) | 1 | 0
Popliteal vein thrombosis (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT02507505/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT02507505/SAP_001.pdf